CLINICAL TRIAL: NCT02586519
Title: Pressure-Sensing Insoles in the Neuropathic Ulcer Treatment Pathway (PINUP): A Randomized Controlled Trial for Active Neuropathic Ulcer Treatment
Brief Title: Pressure-Sensing Insoles in the Neuropathic Ulcer Treatment Pathway
Acronym: PINUP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: During the unavoidable gap resulting from the global pandemic, the technologies being used in this study have significantly improved and it is no longer optimal to provide patients with the old technology when improved technology is available.
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Karim Manji, Clinical Lecturer, Department of Surgery, University of Calgary, Cumming School of Medicine, Diabetic Foot & Limb Preservation Centre Peter Lougheed Centre, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PINUP
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Diabetes; Diabetes Complications; Neuropathy; Peripheral Neuropathy; Diabetic Foot Ulcer
Keywords: wearable technology; Orpyx; SurroSense Rx; smart insole; TCC; total contact cast; insole; removable cast walker; RCW
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Complications; Peripheral Nervous System Diseases; Diabetic Foot

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active SurroSense Rx System + RCW (Experimental): Patients randomized to the experimental group will be fitted with an active (alerting) version of the SurroSense R® smart insole System. This device will be placed in the RCW, underneath the liner. The device tab will be fed up the instep, through a hole in the liner, and affixed to the dorsum of the RCW by way of a tie.
  Interventions: Device: SurroSense Rx System
- Inactive SurroSense Rx System + RCW (Sham Comparator): Patients randomized to this group will be fitted with an inactive (non-alerting) version of the device in an identical fashion.
  Interventions: Device: SurroSense Rx System
- Inactive SurroSense Rx System + iTCC (Sham Comparator): Patients in this group will be fitted with an inactive (non-alerting) version of the device in an identical fashion. The RCW will be further secured using a device specific tie such that it acts as an iTCC.
  Interventions: Device: SurroSense Rx System

INTERVENTIONS:
Device: SurroSense Rx System — The SurroSense Rx system (Orpyx Medical Technologies Inc., Calgary, AB) is a smart insole system designed to aid in the prevention of plantar pressure ulceration and re-ulceration, and the treatment of active ulcers in neuropathic patients. It comprises two pressure-sensing inserts and a smartwatch display device. The device alerts the user when "safe" pressure and time thresholds have been exceeded so that on-demand offloading can occur.
  Other Names: SurroSense Rx Smart Insole System

SUMMARY:
Diabetic foot ulceration (DFU) is a common complication with a 25% lifetime risk in patients with diabetes. While most of these ulcers can be treated successfully on an outpatient basis, some will persist and become infected. Nearly one fifth of patients with lower-extremity diabetic ulcers will require amputation of the affected limb, resulting in staggering costs for both the patient and the healthcare system. Therapies that promote rapid and complete healing and reduce the need for expensive surgical procedures impact these costs substantially.

The standard of care for the treatment of diabetic foot ulcers is the removable cast walker (RCW). RCW use has demonstrated plantar pressure reduction yet is typically perceived as having compliance issues due to its removable nature. In addressing this limitation, a modified version of the RCW has been developed by wrapping it in a layer of cohesive or plaster bandage. This technique has been termed the "instant" total contact cast (iTCC) derived from the seldom-used, gold standard treatment, the total contact cast (TCC). While ease of application and potential clinical equivalence are clear benefits, the iTCC carries disadvantages on account of its irremovability. For example, frequent dressing changes impractical, yet may be necessary for complex wound care. The goal of this research is to continue inquiry and innovation in this most basic aspect of care, whilst addressing the limitations of past research and failures in this domain.

The investigators propose examining the capability of the SurroSense Rx® smart insole and smartwatch system (Orpyx Medical Technologies Inc., Calgary AB) in managing and monitoring adherence to plantar pressure offloading through alert-based feedback. The insoles are embedded with pressure sensors, which wirelessly communicate with a smartwatch that provides feedback on modifying activity or pressure profile over time. This smartwatch transmits audio, visual, and tactile notifications when excessive pressure-time thresholds under plantar regions of interest have been met. This feedback allows patients to be educated on their plantar pressure, and engages them and their caregivers to manage adherence to offloading. The investigators also propose comparing the healing rates of active neuropathic ulcers using RCWs coupled with the SurroSense Rx® smart insole system to assess whether adjunctive use of the two interventions improves the efficiency of neuropathic ulcer treatment.

DETAILED DESCRIPTION:
Pressure offloading is the lynchpin of neuropathic ulcer care. Multiple methods of statically reducing pressure have been employed, with various degrees of success, in the ulcer care continuum. Traditional offloading interventions redistribute the load on the plantar surface, and include: non-removable devices (total contact casts, removable walkers rendered non-removable, and cast shoes), and removable devices (walkers, forefoot offloading shoes, half shoes, bivalve total contact casts, and therapeutic shoes)1,2,3.

A Cochrane Review on the use of offloading in the treatment of uncomplicated neuropathic plantar ulcers gives the efficacy of each device type in terms of percentage of ulcers healed and time required for healing4. The total contact cast has been found to be more effective than removable devices in many randomized controlled trials, for both the percentage of neuropathic ulcers healed and the time required for healing5,6,7. Ninety-two percent of neuropathic ulcers healed in an average of 6 weeks8. Removable walkers made non-removable may be as effective as total contact casts9,10,11. The effectiveness of forefoot offloading shoes, half-shoes, and cast shoes in the healing of neuropathic forefoot ulcers needs to be confirmed by prospective trials12. The lower efficacy of prescribed removable devices could be attributable to a lower adherence to recommended use13.

The effectiveness of offloading interventions is intimately linked to the skin reperfusion that is seen when persistent external pressure is alleviated. Key modifiable parameters in mitigating tissue damage to the neuropathic foot are pressure and time. Kosiak reported in 1959 that "microscopic pathologic changes were noted in tissues subjected to as little as 60 mmHg for only one hour"14,15. More recently, exposures from 15 min to one hour at pressures greater than 240 mmHg, and from two hours or more at pressures greater than 67 mmHg, were found to cause cell death in rat muscle tissue16. Despite this, there is limited information regarding the efficacy of interventions aimed at preventing pressure ulcers; a comprehensive review of the literature did not find enough evidence to recommend a repositioning frequency17. A consensus document from an international review on pressure ulcer prevention states that "patients confined to wheelchairs should be taught to reposition every 15 minutes"18.

While established pressure offloading interventions are able to statically reduce pressure on the active ulcer, they provide no dynamic relief of pressure. Since neuropathy is characterized by a loss of protective sensation (LOPS), the patient is often unaware of sustained pressure on a specific anatomic region over time. Even with static offloading instruments, it is conceivable that critical pressure and time thresholds can be dynamically exceeded without the patient's knowledge or ability to address the problem.

Taken together, the literature provides support for the development of a system that monitors pressure over time at key locations, and provides alert-based feedback to guide as-needed, patient-based offloading for use in patients with active ulceration.

The SurroSense Rx system (Orpyx Medical Technologies Inc., Calgary, AB) is a patent pending (US Publication #20120109013 and PCT WO/2012/055029) footwear system designed to aid in the prevention of plantar pressure ulceration and re-ulceration and the treatment of active ulcers in neuropathic patients. It comprises two pressure-sensing inserts and a smartwatch display device. The device alerts the user when "safe" pressure and time thresholds have been exceeded; the current thresholds are based on the general clinical understanding of pressure ulcer formation, which indicates that a conservative threshold would be >30-50mmHg for >15 minutes. For a review of the literature, please refer to Appendix 4. As more plantar pressure and outcome data are collected over time, these thresholds may be modified for future iterations of the product. These thresholds will be kept constant for the duration of the study in question. The device measures plantar pressures at discrete points corresponding to bony prominences that would be considered to be at higher risk for ulceration: the first metatarsal head (1), the lateral metatarsal heads (2), the great toe (1), the lateral toes (1), the lateral foot (2), and the heel (1). These areas were selected based on the inherent high risk of neuropathic ulceration at these anatomic locations. This data is tracked, with analysis being performed on those that have been collected over the last 15 minutes. If > 95% of the measurements taken by a pressure sensor over a 15-minute scanning window exceed 30-50 mmHg, an alert is sent to the user via the smartwatch to guide them to appropriately offload that area.

The proof of concept of the designed platform as a supplement in the management of the diabetic foot ulcer (DFU) will be assessed in the context of a randomized clinical trial (RCT) pilot. Our hypotheses are that the proposed technology will:

1. Accelerate the wound healing process (i.e. success of complete wound healing within 16 weeks, time to heal, rate of wound size change, and complication rate);
2. Improve adherence with RCW use (measured in hours of use per day); and
3. Improve offloading (i.e. in terms of pressure-time intervals).
4. Upon wound closure, prevent the incidence of plantar ulcer recurrence.

Eligible subjects will be randomized to the Experimental Arm, Control Arm A or Control Arm B (25 per arm). The experimental group will be provided with an active (alerting) SurroSense Rx® device fitted into a standardized RCW* (Rebound® Diabetic Walker, Össur, Iceland). Control Group A will be provided with an inactive (non-alerting) version of the SurroSense Rx® device fitted into a standardized RCW. Control Group B will be provided with an inactive version of the SurroSense Rx® device fitted into a standardized RCW and secured with a device-specific tie; this will act as an iTCC device for the purposes of this trial. Patients in all arms will be provided with a New Balance 928 shoe to wear on their contralateral foot so as to ensure optimal device performance. All patients will be assessed at baseline and every week until successful wound healing or 16 weeks, whichever comes first. Following wound resolution, patients will be followed with their assigned device, being used in a pair of New Balance 928 shoes to be provided to the patient, for 6 months for ulcer recurrence. After 6 months, the device will be discontinued, at which time the patients will be followed for an additional 12 months for further ulcer recurrence. Should a patient's wound remain unresolved after 16 weeks, they will continue using their assigned device into the subsequent 6-month period. If wound resolution occurs during this 6-month period, patients will switch to the New Balance 928 shoes for the remainder of the period; however, if wound resolution does not occur during this time, the patient will be withdrawn from the study prior to the commencement of the subsequent 12-month observation period. For all research subjects wearing the SurroSense Rx®, the device will measure plantar pressure and adherence to prescribed offloading. All groups will be fit with Jawbone UP Activity Trackers (or an equivalent activity tracker) so as to monitor their activity throughout the study.

*The removable Rebound® Diabetic Walker insole is heat-moldable: it can be heated (3 minutes at 110°C/230°F) and formed to the patients' foot (the patient stands in socks on the heated insole for 1 minute - then the hexagons should be removed as appropriate). This method should improve the weight distribution of the plantar foot and provide better offloading at the ulcer sites, and is recommended for optimal treatment.

Primary aims of the study:

* This pilot study will investigate the efficacy of the SurroSense Rx® system in expediting the healing of active neuropathic ulcers in terms of rate of wound area reduction.
* It will also investigate the system's potential to improve healing rates in the treatment of active neuropathic ulcers using the more practical RCWs.
* It will also investigate the system's potential to prevent recurrent ulceration post ulcer resolution. To achieve this, following wound resolution, patients will be followed for 18 months (the first 6 months with their assigned device) to monitor for ulcer recurrence.

Secondary aims of the study:

* Compare complete wound healing at 16 weeks in the experimental versus control groups
* Compare the healing times and rates as a function of the patient's baseline Michigan Neuropathy Screening Instrument (MNSI) and Modified Neuropathy Disability Score (MNDS)19 in the experimental versus control group
* Compare the change in the MNDS over the course of the study
* Performance of a cost-effectiveness analysis of the experimental versus control group's methods of treating diabetic ulcers
* Elucidate pressure data and adherence parameters (activity data-including step count and type of activity, peak pressures, number of alerts, measures of central tendency for time to offload, areas of alert generation, hours of use per day) for all patients, and compare those data for patients in the experimental versus control groups
* Compare area of ulceration to areas of SurroSense Rx® device alert generation (active devices) or would-be alert generation (inactive devices)
* Compare pressure data and adherence parameters (activity data-including step count and type of activity, peak pressures, number of alerts, measures of central tendency for time to offload, areas of alert generation, hours of use per day) to MNSI and MNDS Scales
* Examine the ability of pressure data and adherence parameters to predict healing
* Comparison of complication rates in the experimental versus control groups

ELIGIBILITY:
Inclusion Criteria:

* Diabetes (according to AAFP diagnostic criteria )
* Presence of neuropathy with Loss of Protective Sensation (LOPS), as defined by any loss of sensation as per the assessments included in the Modified Neuropathy Disability Score (MNDS)
* Active plantar diabetic foot ulcer (Grade 1A, according to the University of Texas Wound Classification System , )

  * A minimum size ulcer ≥0.5cm2 and ≤ 12 cm2 post debridement at time of randomization
  * If the subject has more than one ulcer, they should be identified and at least 2 cm apart
* Age >18
* At least one palpable foot pulse
* Ability to understand all of the study requirements
* Life expectancy greater than the duration of the study
* Subject or responsible caregiver is willing and able to maintain the required offloading (as applicable for the location of the ulcer) and applicable dressing changes
* Doppler Ultrasound positive for at least one pedal pulse in each foot

Exclusion Criteria:

* Weight > 400 lb (182 kg)
* Uncorrected visual impairment
* Active Infection
* Non-plantar ulcers on the ankle, posterior heel, or other location
* More than one active plantar ulcer
* Presence of severe ischemia (any of: absence of foot pulses, Ankle Brachial Index 0.6 > [ABI] > 1.2, capillary refill time > 5 seconds; see Appendix 3)
* Current participation in another clinical investigation of a medical device or a drug; or has participated in such a study within 30 days prior to this study
* Current smokers
* Active abuse of alcohol

  o Subject has a history of any of the following intercurrent illnesses or conditions that would compromise the safety of the subject or the normal healing process:
* End-stage renal disease
* Immunosuppression
* Severe malnutrition
* Liver disease
* Aplastic anemia
* Scleroderma
* Acquired immune deficiency disease (AIDS) or HIV positive
* Connective tissue disorder
* Exacerbation of sickle cell anemia
* Active Charcot foot
* Excessive lymphedema
* Osteomyelitis and gangrene
* Subjects with ulcers secondary to a disease other than diabetes (e.g. vasculitis, neoplasms or haematological disorders)

  o At the end of the run-in period and prior to randomization, the subject be excluded if the following conditions are not met:
* Subject does not continue to meet the entrance criteria (inclusion and exclusion)
* The size of the study ulcer, following debridement, has decreased by more than 30% from the baseline assessment measured at screening.
* Abnormal toe and/or ankle range of motion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Rate of Wound Closure | 12 Weeks
  Rate of Wound Closure (mm2 per day)
Rate of Wound Resolution | 12 weeks
  Rate of Wound Closure (Complete) over first 12 weeks

SECONDARY OUTCOMES:
Recurrence of Ulcer | 6 months
  Rate of ulcer recurrence in 6 months post complete wound closure (epithelialization)
Cost Utility | Wound Healing Period (up to 12 weeks) + 6 Months Post-Wound Closure
  Cost of care over assessed period
Activity | Wound Healing Period (up to 12 weeks) + 6 Months Post-Wound Closure
  Change in activity (step count) over time period of assessment
Complication Rates | Wound Healing Period (up to 12 weeks)
  Requirement for antibiotics and/or surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Karim Manji, DPM, AACFAS, Principal Investigator — University of Calgary
Locations (1):
- Zivot Limb Preservation Centre- Peter Lougheed Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavanagh PR, Bus SA. Off-loading the diabetic foot for ulcer prevention and healing. J Vasc Surg. 2010 Sep;52(3 Suppl):37S-43S. doi: 10.1016/j.jvs.2010.06.007. PMID 20804932
- [Background] Bus SA, Valk GD, van Deursen RW, Armstrong DG, Caravaggi C, Hlavacek P, Bakker K, Cavanagh PR. The effectiveness of footwear and offloading interventions to prevent and heal foot ulcers and reduce plantar pressure in diabetes: a systematic review. Diabetes Metab Res Rev. 2008 May-Jun;24 Suppl 1:S162-80. doi: 10.1002/dmrr.850. PMID 18442178
- [Background] Bus SA. Priorities in offloading the diabetic foot. Diabetes Metab Res Rev. 2012 Feb;28 Suppl 1:54-9. doi: 10.1002/dmrr.2240. PMID 22271724
- [Background] Lewis J, Lipp A. Pressure-relieving interventions for treating diabetic foot ulcers. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD002302. doi: 10.1002/14651858.CD002302.pub2. PMID 23440787
- [Background] KOSIAK M. Etiology and pathology of ischemic ulcers. Arch Phys Med Rehabil. 1959 Feb;40(2):62-9. No abstract available. PMID 13618101
- [Background] Linder-Ganz E, Engelberg S, Scheinowitz M, Gefen A. Pressure-time cell death threshold for albino rat skeletal muscles as related to pressure sore biomechanics. J Biomech. 2006;39(14):2725-32. doi: 10.1016/j.jbiomech.2005.08.010. Epub 2005 Sep 30. PMID 16199045
- [Background] Reddy M, Gill SS, Rochon PA. Preventing pressure ulcers: a systematic review. JAMA. 2006 Aug 23;296(8):974-84. doi: 10.1001/jama.296.8.974. PMID 16926357
- [Background] Chawla A, Bhasin G, Chawla R, "Validation Of Neuropathy Symptoms Score (NSS) And Neuropathy Disability Score (NDS ) In The Clinical Diagnosis Of Peripheral Neuropathy In Middle Aged People With Diabetes." The Internet Journal of Family Practice; 12(1).
- [Background] Armstrong DG, Lavery LA, Harkless LB. Validation of a diabetic wound classification system. The contribution of depth, infection, and ischemia to risk of amputation. Diabetes Care. 1998 May;21(5):855-9. doi: 10.2337/diacare.21.5.855. PMID 9589255
- [Background] Lavery LA, Armstrong DG, Harkless LB. Classification of diabetic foot wounds. J Foot Ankle Surg. 1996 Nov-Dec;35(6):528-31. doi: 10.1016/s1067-2516(96)80125-6. PMID 8986890
- [Background] Mueller MJ, Diamond JE, Sinacore DR, Delitto A, Blair VP 3rd, Drury DA, Rose SJ. Total contact casting in treatment of diabetic plantar ulcers. Controlled clinical trial. Diabetes Care. 1989 Jun;12(6):384-8. doi: 10.2337/diacare.12.6.384. PMID 2659299
- [Background] Ganguly S, Chakraborty K, Mandal PK, Ballav A, Choudhury S, Bagchi S, Mukherjee S. A comparative study between total contact casting and conventional dressings in the non-surgical management of diabetic plantar foot ulcers. J Indian Med Assoc. 2008 Apr;106(4):237-9, 244. PMID 18828342
- [Background] Armstrong DG, Lavery LA, Wu S, Boulton AJ. Evaluation of removable and irremovable cast walkers in the healing of diabetic foot wounds: a randomized controlled trial. Diabetes Care. 2005 Mar;28(3):551-4. doi: 10.2337/diacare.28.3.551. PMID 15735186
- [Background] Ahn C, Salcido RS. Advances in wound photography and assessment methods. Adv Skin Wound Care. 2008 Feb;21(2):85-93; quiz 94-5. doi: 10.1097/01.ASW.0000305411.58350.7d. PMID 18349736
- [Background] Thomas GB, Finney RL. Calculus and Analytic Geometry. 9th ed. Reading, MA: Addison Wesley; 1995.